CLINICAL TRIAL: NCT02721966
Title: MAXIMISE (Managing AXIal Manifestations in PsorIatic Arthritis With SEcukinumab), a Randomized, Double-blind, Placebo-controlled, Multicenter, 52-week Study to Assess the Efficacy and Safety of Secukinumab 150 mg or 300 mg s.c. in Participants With Active Psoriatic Arthritis and Axial Skeleton Involvement Who Have Inadequate Response to Non-steroidal Anti-inflammatory Drugs (NSAIDs)
Brief Title: Study of the Efficacy and Safety of Secukinumab in Participants With Active Psoriatic Arthritis With Axial Skeleton Involvement
Acronym: MAXIMISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F3302; 2016-000814-31 (EudraCT Number)
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Axial Psoratic Arthritis
Keywords: Assessment of spondyloarthritis international society; ASAS; axial; Psoriatic Arthritis; PsA; Magnetic resonance imaging; MRI
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: 498 patients were randomized in this Phase 3b trial. 5 (of 503) were mis-randomized, i.e. received randomization number but never received study medication.
  This was a 52-week, randomized, double-blind, double-dummy, placebo-controlled, multicenter study to assess the efficacy of secukinumab 150 mg or 300 mg in patients with AxPsA who had an inadequate response to NSAIDs. The study had 2 treatment periods; a placebo-controlled period from Baseline to Week 12 followed by an active treatment period from Week 12 to Week 52.
  At Week 12, patients randomized to placebo at Baseline were re-randomized (1:1) to active treatment with secukinumab 150 mg or secukinumab 300 mg.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AIN457 150mg (Experimental): Secukinumab dose amount 1 sc injection weekly for 4 weeks followed by Secukinumab dosage amount 1 sc injection every 4 weeks for remaining 44 weeks
  Interventions: Biological: Secukinumab
- AIN457 300mg (Experimental): Secukinumab dose amount 2 sc injection weekly for 4 weeks followed by Secukinumab dosage amount 2 sc injection every 4 weeks for remaining 44 weeks
  Interventions: Biological: Secukinumab
- AIN457 Placebo (Placebo Comparator): Placebo sc injection weekly for 4 weeks and at week 8, followed by Secukinumab 150 mg or 300 mg sc injection every 4 week for remaining 40 weeks.
  Interventions: Biological: Secukinumab; Drug: Secukinumab and Placebo

INTERVENTIONS:
Biological: Secukinumab — Anti IL-17a monoclonal antibody
  Other Names: AIN457
Drug: Secukinumab and Placebo — Placebo matching AIN457
  Arms: AIN457 Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of secukinumab 150 mg or 300 mg in the management of axial manifestations in PsA patients who have failed to respond to at least 2 non-steroidal anti-inflammatory drugs (NSAIDs) over a 4-week period, according to assessment of spondyloarthritis international society (ASAS) recommendations for the treatment of axial spondyloarthritis (AxSpA).

DETAILED DESCRIPTION:
In the anlalysis (CSR), there are 498 patients, as 5 patients were mis-randomized, i.e. had randomization number but did never take study medication. So there were 498 participants, and not 503

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed
* Diagnosis of psoriatic arthritis classified by Classification criteria for psoriatic arthritis (CASPAR) criteria
* Active spinal disease defined by Bath ankylosing spondylitis disease activity index (BASDAI) score ≥ 4
* Spinal Pain visual analog scale (VAS) ≥ 40 (on a VAS 100 scale)
* Inadequate Response to at least 2 non-steroidal anti-inflammatory drugs over a 4 weeks period

Exclusion Criteria:

* History of exposure to other IL-17 or IL-23 inhibitor biologic drug
* History of exposure to previous biologic disease modifying anti-rheumatic drugs (DMARDs) (Tumor necrosis factor (TNF) blockers or Ustekinumab)
* Current treatment with disease modifying anti-rheumatic drugs (DMARDs) other than Methotrexate
* Subjects taking high potency opioid analgesics (e.g. methadone, hydromorphone, morphine)
* Chest X-ray or chest magnetic resonance imaging (MRI) with evidence of ongoing infectious or malignant process, obtained within 3 months prior to screening and evaluated by a qualified physician

Other protocol-defined inclusion and exclusion criteria may have applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (84):
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Bulgaria (2):
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sofia
- Czechia (4):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Bruntál
  - Novartis Investigative Site, Plzen-Bory
  - Novartis Investigative Site, Uherské Hradiště
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Finland (2):
  - Novartis Investigative Site, Kuopio
  - Novartis Investigative Site, Kuovola
- France (6):
  - Novartis Investigative Site, Strasbourg, Cedex
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Cottbus
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Magdeburg
- Novartis Investigative Site, Athens, Greece
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Hévíz
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Veszprém
- Novartis Investigative Site, Dublin, Ireland
- Israel (4):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Bologna
- Poland (6):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Piotrkow Trybunalski
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Romania (2):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
- Russia (9):
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Khanty-Mansiysk
  - Novartis Investigative Site, Kursk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Orenburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Yaroslavl
- Spain (15):
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Terrassa, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Lugo, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Las Palmas de Gran Canaria, Las Palmas de G.C
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Pontevedra
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Vitoria-Gasteiz
- Switzerland (4):
  - Novartis Investigative Site, Fribourg, CH
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Zurich
- United Kingdom (9):
  - Novartis Investigative Site, Devon, Barnstaple
  - Novartis Investigative Site, Basingstoke, Hampshire
  - Novartis Investigative Site, Maidstone, Kent
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, Wigan
  - Novartis Investigative Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Baraliakos X, Pournara E, Coates LC, Navarro-Compan V, Blanco R, O'Brien E, Schulz B, Landewe R. Magnetic resonance imaging characteristics in patients with psoriatic arthritis and axial manifestations from the MAXIMISE cohort. Rheumatology (Oxford). 2024 Jan 4;63(1):85-92. doi: 10.1093/rheumatology/kead162. PMID 37094184
- [Derived] Baraliakos X, Gossec L, Pournara E, Jeka S, Mera-Varela A, D'Angelo S, Schulz B, Rissler M, Nagar K, Perella C, Coates LC. Secukinumab in patients with psoriatic arthritis and axial manifestations: results from the double-blind, randomised, phase 3 MAXIMISE trial. Ann Rheum Dis. 2021 May;80(5):582-590. doi: 10.1136/annrheumdis-2020-218808. Epub 2020 Dec 17. PMID 33334727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 503 participants completed the screening period; and the randomized set consists of 498 patients because 5 participants were misrandomized
Pre-assignment Details: 95.6% of those randomized completed period 1 and moved on to period 2; and the 85.3% completed treatment period 2.
Groups:
- AIN457 300mg: Secukinumab 300 mg sc injections at baseline and weekly until 4 weeks followed by Secukinumab 300 mg injections every 4 weeks between week 8 and week 48
- AIN457 150mg: Secukinumab 150 mg sc injections at baseline and weekly until 4 weeks followed by Secukinumab 150 mg injections every 4 weeks between week 8 and week 48
- Placebo AIN457 300 mg: Placebo sc injection weekly for 4 weeks and at week 8, followed by Secukinumab 300 mg sc injection every 4 week for remaining 40 weeks.
- Placebo AIN457 150 mg: Placebo sc injection weekly for 4 weeks and at week 8, followed by Secukinumab 150 mg sc injection every 4 week for remaining 40 weeks.
- Placebo: Placebo sc injections at baseline and weekly until Week 8
Period: Overall Study
Arm/Group | AIN457 300mg | AIN457 150mg | Placebo AIN457 300 mg | Placebo AIN457 150 mg | Placebo
Started (Randomized) | 167 | 165 | 81 | 80 | 5
Completed Period 1 & Went to Period 2 | 162 | 153 | 81 | 80 | 0
Completed (Completed treatment period 2) | 138 | 142 | 72 | 73 | 0
Not Completed | 29 | 23 | 9 | 7 | 5
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 2 | 3 | 7 | 0
Not completed — Adverse Event | 4 | 4 | 3 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 7 | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Did not continue to period 2 | 5 | 12 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Randomized set: All participants randomized to AIN457 300 mg/150 mg or Placebo.
Groups:
- Placebo AIN457: Placebo sc. injections at baseline and weekly until Week 4, then at Week 8 and followed by Secukinumab 300 mg or 150 mg injections every 4 weeks between week 12 and week 48
- Total: Total of all reporting groups
Arm/Group | AIN457 300mg | AIN457 150mg | Placebo AIN457 | Total
Number analyzed (Participants) | 167 | 165 | 166 | 498
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 159 | 156 | 157 | 472
  >=65 years | 8 | 9 | 9 | 26
Age, Customized [Count of Participants; unit: Participants] — age in years
  Participants
    <45 years old | 77 | 65 | 72 | 214
    >=45 years old | 90 | 100 | 94 | 284
Sex: Female, Male [Count of Participants; unit: Participants] — Of 498 participants, 50.6% of participants were female, and 49.4% were male
  Participants
    Female | 90 | 84 | 78 | 252
    Male | 77 | 81 | 88 | 246
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Of 498 participants, , 0.2% of participants were Black, 0.4% were Asian, 97.4% were White, and 2.0% were Unknown
  Participants
    Black | 1 | 0 | 0 | 1
    Asian | 0 | 0 | 2 | 2
    White | 162 | 159 | 164 | 485
    Unknown | 4 | 6 | 0 | 10
Race/Ethnicity, Customized [Number; unit: Participants] — Of 498 participants, 5.0% of participants were Hispanic or Latino, and 85.3% were not.
  Participants
    Hispanic or Latino | 6 | 10 | 9 | 25
    Not Hispanic or Latino | 139 | 140 | 146 | 425
    Not reported | 17 | 10 | 8 | 35
    Unknown | 5 | 5 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response to Treatment (300 mg AIN457) as Assessed by the ASAS20 Criteria at Week 12
Description: Purpose of this measure: was to demonstrate that secukinumab 150 mg s.c. is superior to placebo in the achievement of ASAS 20 response at Week 12 after superiority of 300 mg was established
  ASAS20 was defined as an improvement of ≥20% and absolute improvement of ≥10 unit (0-100 mm VAS) from baseline in ≥3 of the following 4 domains (and absence of deterioration in any domain): patient's global assessment of disease activity (PTGA), pain assessment (total pain score), Bath Ankylosing Spondylitis Functional Index (BASFI), and clinical inflammation (mean of 2 morning stiffness-related scores on the BASDAI)
Time Frame: at week 12
Population: Full analysis set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo AIN457
Number analyzed (Participants) | 157 | 164 | 164
percentage of participants | 66.3 [58.4 to 73.3] | 62.9 [55.2 to 70.0] | 31.2 [24.6 to 38.7]
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo AIN457; Up to week 12, all participants in the group "placebo AIN457" took placebo only; Test type: Superiority; p < .0001, Regression, Logistic; 95% confidence interval for odds ratio; Odds Ratio (OR) = 4.37, 95% CI 2-sided [2.72 to 7.01]
Statistical Analysis 2: Comparison: AIN457 300mg vs Placebo AIN457; Up to week 12, all participants in the group "placebo AIN457" took placebo only; Test type: Superiority; p < .0001, Regression, Logistic; 95% confidence interval for odds ratio; Odds Ratio (OR) = 3.83, 95% CI 2-sided [2.41 to 6.10]

2. Secondary Outcome: Percentage of Participants With Response to Treatment (150 mg AIN457) as Assessed by the ASAS20 Criteria at Week 12
Description: Purpose of this key secondary measure: was to demonstrate that secukinumab 150 mg s.c. is superior to placebo in the achievement of ASAS 20 response at Week 12 after superiority of 300 mg was established. 300mg and 150mg are presented side by side for clarity; and to align with protocol. 300mg data is for Primary outcome; and 150mg data is for key secondary outcome
  ASAS20 was defined as an improvement of ≥20% and absolute improvement of ≥10 unit (0-100 mm VAS) from baseline in ≥3 of the following 4 domains (and absence of deterioration in any domain): patient's global assessment of disease activity (PTGA), pain assessment (total pain score), Bath Ankylosing Spondylitis Functional Index (BASFI), and clinical inflammation (mean of 2 morning stiffness-related scores on the BASDAI)
Time Frame: at week 12
Population: Full analysis set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo AIN457
Number analyzed (Participants) | 157 | 164 | 164
percentage of participants | 66.3 [58.4 to 73.3] | 62.9 [55.2 to 70.0] | 31.2 [24.6 to 38.7]
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo AIN457; Up to week 12, all participants in the group "placebo AIN457" took placebo only; Test type: Superiority; p < .0001, Regression, Logistic; 95% confidence interval for odds ratio; Odds Ratio (OR) = 4.37, 95% CI 2-sided [2.72 to 7.01]

3. Secondary Outcome: Percentage of Participants With Response to Treatment (150 mg/300 mg AIN457) as Assessed by the ASAS40 Criteria at Week 12
Description: Proportion of patients with response to treatment as assessed by the Assessment of spondyloarthritis international society (ASAS) 40 criteria at week 12.
  ASAS40 was defined as an improvement of ≥40% and absolute improvement of ≥20 unit (0-100 mm VAS) from baseline in ≥3 of the following 4 domains (and absence of deterioration in any domain): patient's global assessment of disease activity (PTGA), pain assessment (total pain score), Bath Ankylosing Spondylitis Functional Index (BASFI), and clinical inflammation (mean of 2 morning stiffness-related scores on the BASDAI)
Time Frame: at week 12
Population: Full analysis set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo AIN457
Number analyzed (Participants) | 157 | 164 | 164
percentage of participants | 39.5 [32.1 to 47.4] | 43.6 [36.2 to 51.3] | 12.2 [7.8 to 18.4]
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo AIN457; Test type: Superiority; p < .0001, Regression, Logistic; 95% confidence interval for odds ratio; Odds Ratio (OR) = 4.71, 95% CI 2-sided [2.67 to 8.33]; Odds ratio, 95% CI for odds ratio, and p-value are from a logistic regression model with treatment (3 treatment groups), methotrexate usage status (yes, no) as explanatory variables
Statistical Analysis 2: Comparison: AIN457 300mg vs Placebo AIN457; Test type: Superiority; p < .0001, Regression, Logistic; 95% confidence interval for odds ratio; Odds Ratio (OR) = 5.61, 95% CI 2-sided [3.20 to 9.84]; [other analysis details as in outcome 3, analysis 1]

4. Secondary Outcome: Percentage of Participants With Response to Treatment as Assessed by BASDAI50 at Week 12
Description: Bath ankylosing spondylitis disease activity index (BASDAI) 50 response
  BASDAI 50 response is defined as at least 50% improvement (decrease) in total BASDAI score.
Time Frame: at week 12
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of particiapnts
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo AIN457
Number analyzed (Participants) | 157 | 164 | 164
percentage of particiapnts | 32.7 [25.8 to 40.5] | 37.4 [30.1 to 45.4] | 9.8 [5.9 to 15.6]
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo AIN457; Up to week 12, all participants in the group "placebo AIN457" took placebo only; Test type: Superiority; p < .0001, Regression, Logistic; 95% confidence interval for odds ratio; Odds Ratio (OR) = 4.50, 95% CI 2-sided [2.43 to 8.33]; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: AIN457 300mg vs Placebo AIN457; Up to week 12, all participants in the group "placebo AIN457" took placebo only; Test type: Superiority; p < .0001, Regression, Logistic; 95% confidence interval for odds ratio; Odds Ratio (OR) = 5.57, 95% CI 2-sided [3.04 to 10.21]; [other analysis details as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline in Spinal Pain Visual Analog Scale (VAS) - Pain at Any Time
Description: Change from baseline in Spinal pain visual analog scale (VAS) at week 12
  VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom,pain,health) orientated from the left (worst) to the right (best).
  VAS measures pain and stress for on a horizontal line of 100 mm, ranging from very low (0) to very high (100).
Time Frame: at baseline, at week 12
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo AIN457
Number analyzed (Participants) | 157 | 164 | 164
scores on a scale | -28.5 (1.88) | -26.5 (1.84) | -13.6 (1.83)
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo AIN457; Test type: Superiority; p < .0001, ANCOVA; LS Mean of Treatment Difference = -14.9, 95% CI 2-sided [-20.0 to -9.7], Standard Error of Mean 2.62; Least squares (LS) mean, LS mean treatment difference, 95% confidence interval (CI) for treatment difference, and p-value are from MMRM (mixed model for repeated measures) with treatment group, visit, treatment*visit, baseline*visit and concomitant MTX intake status, as factors and baseline measurement in VAS as continuous covariate
Statistical Analysis 2: Comparison: AIN457 300mg vs Placebo AIN457; Test type: Superiority; p < .0001, ANCOVA; LS Mean of Treatment Difference = -12.9, 95% CI 2-sided [-18.0 to -7.8], Standard Error of Mean 2.59; [other analysis details as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline in Spinal Pain Visual Analog Scale (VAS) - Pain at Night
Description: as for outcome 5
Time Frame: at baseline, at week 12
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo AIN457
Number analyzed (Participants) | 157 | 164 | 164
scores on a scale | -30.3 (1.95) | -30.2 (1.90) | -15.2 (1.89)
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo AIN457; Up to week 12, all participants in the group "placebo AIN457" took placebo only; Test type: Superiority; p < .0001, ANCOVA; LS Mean of Treatment Difference = -15.1, 95% CI 2-sided [-20.4 to -9.7], Standard Error of Mean 2.71; [other analysis details as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: AIN457 300mg vs Placebo AIN457; Up to week 12, all participants in the group "placebo AIN457" took placebo only; Test type: Superiority; p < .0001, ANCOVA; LS Mean of Treatment Difference = -15.0, 95% CI 2-sided [-20.3 to -9.8], Standard Error of Mean 2.68; [other analysis details as in outcome 5, analysis 1]

7. Secondary Outcome: Change From Baseline Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index Score at Week 12
Description: The Spondyloarthritis Research Consortium of Canada (SPARCC) enthesitis index score range is 0-16, where 0 is the best outcome, and 16 the worst. The assessor determines whether the site shows tenderness and therefore would count as site with enthesitis. This is done by applying pressure to the site and getting feedback from patient about whether the site is tender.
Time Frame: baseline and week 12
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo AIN457
Number analyzed (Participants) | 157 | 164 | 164
scores on a scale | -2.2 (0.22) | -2.4 (0.21) | -1.7 (0.21)
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo AIN457; Test type: Superiority; p = 0.0971, ANCOVA; LS Mean of Treatment Difference = -0.5, 95% CI 2-sided [-1.1 to 0.1], Standard Error of Mean 0.30; Least squares (LS) mean, LS mean treatment difference, 95% confidence interval (CI) for treatment difference, and p-value are from MMRM (mixed model for repeated measures) with treatment group, visit, treatment*visit, baseline*visit and concomitant MTX intake status, as factors and baseline SPARCC index as continuous covariate
Statistical Analysis 2: Comparison: AIN457 300mg vs Placebo AIN457; Test type: Superiority; p = 0.0207, ANCOVA; LS Mean of Treatment Difference = -0.7, 95% CI 2-sided [-1.3 to -0.1], Standard Error of Mean 0.30; [other analysis details as in outcome 5, analysis 1]

8. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Week 12
Description: The health assessment questionnaire disability index (HAQ-DI) assesses the difficulty a patient has had in the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2-3 items. For each question, level of difficulty is scored from 0 to 3 with 0=no difficulty, 1=some difficulty, 2=much difficulty, and 3=unable to do. The score for each domain is the maximum (worst) score from the items/questions within the domain. Higher score indicates greater disability. Overall score was computed as the sum of the domain scores divided by the number of domains answered. The total possible score ranged from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher overall score indicates greater disability.
Time Frame: baseline and week 12
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo AIN457
Number analyzed (Participants) | 157 | 164 | 164
scores on a scale | -0.330 (0.0360) | -0.389 (0.0353) | -0.155 (0.0351)
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo AIN457; Test type: Superiority; p = 0.0005, ANCOVA; LS Mean of Treatment Difference = -0.175, 95% CI 2-sided [-0.273 to -0.076], Standard Error of Mean 0.0502; Least squares (LS) mean, LS mean treatment difference, 95% confidence interval (CI) for treatment difference, and p-value are from MMRM (mixed model for repeated measures) with treatment group, visit, treatment*visit, baseline*visit and concomitant MTX intake status, as factors and baseline HAQ-DI index as continuous covariate
Statistical Analysis 2: Comparison: AIN457 300mg vs Placebo AIN457; Test type: Superiority; p < .0001, ANCOVA; LS Mean of Treatment Difference = -0.234, 95% CI 2-sided [-0.331 to -0.136], Standard Error of Mean 0.0497; [other analysis details as in outcome 8, analysis 1]

9. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-Fatigue) at Week 12
Description: The FACIT-fatigue scale is a 13-item patient-reported measure of fatigue with a 7-day recall period. Items are scored on a 0 - 4 response scale with anchors ranging from "Not at all" to "Very much so". To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52.
Time Frame: baseline and week 12
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo AIN457
Number analyzed (Participants) | 157 | 164 | 164
scores on a scale | 8.0 (0.72) | 7.6 (0.71) | 4.2 (0.70)
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo AIN457; week 12; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean of Treatment Difference = 3.8, 95% CI 2-sided [1.8 to 5.7], Standard Error of Mean 1.01; Least squares (LS) mean, LS mean treatment difference, 95% confidence interval (CI) for treatment difference, and p-value are from MMRM (mixed model for repeated measures) with treatment group, visit, treatment*visit, baseline*visit and concomitant MTX intake status, as factors and baseline FACIT Fatigue© score as continuous covariate
Statistical Analysis 2: Comparison: AIN457 300mg vs Placebo AIN457; week 12; Test type: Superiority; p = 0.0007, ANCOVA; LS Mean of Treatment Difference = 3.4, 95% CI 2-sided [1.4 to 5.3], Standard Error of Mean 0.99; [other analysis details as in outcome 9, analysis 1]

10. Secondary Outcome: Change From Baseline in Spondyloarthritis International Society (ASAS) Health Index at Week 12
Description: Statistical analysis (using ANCOVA) of change from baseline in spondyloarthritis international society (ASAS) Health Index score by visit - treatment period 1
  ASAS HI is a disease-specific health-index instrument designed to assess the impact of interventions for SpA, including axSpA. The 17-item instrument has scores ranging from 0 (good health) to 17 (poor health). Each item consists of one question that the participant needs to respond to with either "I agree" (score of 1) or "I do not agree" (score of 0). A score of "1" is given where the item is affirmed, indicating adverse health. All item scores are summed to give a total score or index.
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors
Time Frame: baseline and week 12
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo AIN457
Number analyzed (Participants) | 157 | 164 | 164
scores on a scale | -2.9 (0.29) | -2.8 (0.28) | -1.2 (0.28)
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo AIN457; Up to week 12, all participants in the group "placebo AIN457" took placebo only; Test type: Superiority; p < .0001, ANCOVA; LS Mean of Treatment Difference = -1.7, 95% CI 2-sided [-2.5 to -0.9], Standard Error of Mean 0.41; Least squares (LS) mean, LS mean treatment difference, 95% confidence interval (CI) for treatment difference, and p-value are from MMRM (mixed model for repeated measures) with treatment group,visit, treatment*visit, baseline*visit and concomitant MTX intake status, as factors and baseline ASAS health index as continuous covariate
Statistical Analysis 2: Comparison: AIN457 300mg vs Placebo AIN457; Up to week 12, all participants in the group "placebo AIN457" took placebo only; Test type: Superiority; p < .0001, ANCOVA; LS Mean of Treatment Difference = -1.7, 95% CI 2-sided [-2.4 to -0.9], Standard Error of Mean 0.40; [other analysis details as in outcome 10, analysis 1]

11. Secondary Outcome: Percentage of Participants With Response to Treatment as Assessed by the ACR20 Criteria at Week 12
Description: American College of Rheumatology 20% (ACR20) Response at Week 12 is the % of responders with at least 20% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1)Health Assessment Questionnaire-Disability Index (HAQ-DI), 2)C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS)
Time Frame: at week 12
Population: Full analysis set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo AIN457
Number analyzed (Participants) | 157 | 164 | 164
percentage of participants | 56.5 [47.5 to 65.1] | 51.6 [43.4 to 59.8] | 18.5 [13.1 to 25.5]
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo AIN457; Test type: Superiority; p < .0001, Regression, Logistic; 95% confidence interval for odds ratio; Odds Ratio (OR) = 5.74, 95% CI 2-sided [3.31 to 9.95]; Odds ratio, 95% CI for odds ratio, and p-value are from a logistic regression model with treatment (3 treatment groups), methotrexate usage status (yes, no) as explanatory variables. Missing ACR20 response variables were imputed by multiple imputation approach
Statistical Analysis 2: Comparison: AIN457 300mg vs Placebo AIN457; Test type: Superiority; p < .0001, Regression, Logistic; 95% confidence interval for odds ratio; Odds Ratio (OR) = 4.80, 95% CI 2-sided [2.83 to 8.16]; [other analysis details as in outcome 11, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study at week 12
Description: An Adverse Event (AE) is any untoward sign or symptom that occurs during the study treatment
Groups:
- Secukinumab 300 mg: Secukinumab 300 mg sc. injections at baseline and weekly until Week 4 followed by Secukinumab 300 mg injections every 4 weeks between week 8 and week 48 and placebo-switchers to Secukinumab at week 12 onwards
- Secukinumab 150 mg: Secukinumab 150 mg sc. injections at baseline and weekly until Week 4 followed by Secukinumab 150 mg injections every 4 weeks between week 8 and week 48 and placebo-switchers to Secukinumab at week 12 onwards
- Placebo: Placebo sc. injections at baseline and weekly until Week 4, then at Week 8
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/248 | 0/245 | 0/166
Serious Adverse Events (participants affected / at risk) | 14/248 | 14/245 | 4/166
Other Adverse Events (participants affected / at risk) | 116/248 | 108/245 | 47/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (N=248) | Secukinumab 150 mg (N=245) | Placebo (N=166)
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Genitourinary tract infection (Infections and infestations) | 1 | 0 | 0
Peritonsillitis (Infections and infestations) | 1 | 0 | 0
Pyoderma (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (N=248) | Secukinumab 150 mg (N=245) | Placebo (N=166)
Diarrhoea (Gastrointestinal disorders) | 16 | 7 | 4
Vomiting (Gastrointestinal disorders) | 5 | 3 | 1
Fatigue (General disorders) | 6 | 3 | 4
Bronchitis (Infections and infestations) | 11 | 9 | 1
Ear infection (Infections and infestations) | 5 | 2 | 0
Gastroenteritis (Infections and infestations) | 5 | 4 | 2
Nasopharyngitis (Infections and infestations) | 34 | 22 | 11
Pharyngitis (Infections and infestations) | 7 | 13 | 5
Rhinitis (Infections and infestations) | 9 | 5 | 0
Sinusitis (Infections and infestations) | 4 | 6 | 0
Tonsillitis (Infections and infestations) | 7 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 12 | 14 | 5
Urinary tract infection (Infections and infestations) | 8 | 11 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 6 | 1
Blood creatinine increased (Investigations) | 8 | 6 | 0
Hepatic enzyme increased (Investigations) | 5 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 7 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 6 | 6
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 4 | 7 | 1
Headache (Nervous system disorders) | 7 | 7 | 6
Sciatica (Nervous system disorders) | 1 | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 9 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 5 | 6 | 2
Hypertension (Vascular disorders) | 4 | 10 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Publications from a single-site are postponed until publication of the pooled clinical trial data (i.e., data from all sites) or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT02721966/SAP_001.pdf
  • Study Protocol (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT02721966/Prot_002.pdf